CLINICAL TRIAL: NCT01254214
Title: Mindfulness for Symptom Reduction: A Transplant Candidate Study in Program Grant Studies of Organ Transplantation in Animals and Man 2P01 DK013083
Brief Title: Journeys to Wellness: A Transplant Candidate Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0907S70361; 2P01DK013083 (NIH)
Record Dates: First submitted 2010-09-27; First posted 2010-12-06 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: End-stage Renal Disease
Keywords: Mindfulness; Quality of life; Transplantation; Renal disease
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases | interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tMBSR (Experimental): telephone-adapted Mindfulness Based Stress Reduction (tMBSR) is an 8-week program of training in mindfulness meditation consisting of two in-person group meetings and 6 conference calls, led by a trained meditation teacher.
  Interventions: Behavioral: tMBSR
- Support Group (Active Comparator): The Support Group is a group intervention led by a trained facilitator and designed to match the intervention for time, attention and social support
  Interventions: Behavioral: Support group

INTERVENTIONS:
Behavioral: tMBSR — MBSR is an 8-week program of mindfulness meditation and gentle Hatha yoga, taught in a class of up to 30 participants. The telephone-adapted MBSR program (tMBSR) begins with a 5 hour-day workshop to introduce the techniques, followed by 6 weekly 1 ½ hour group teleconferences with the teacher to discuss the class's experiences with meditation practice, and ends with a 5 hour retreat in week 8.
  Other Names: None applicable
  Arms: tMBSR
Behavioral: Support group — The attention control consists of a support group emphasizing communication skills and selecting resources. It includes two 90 minute in-person workshops and 6 1-hour teleconference calls. An experienced facilitator emphasizes communication skills and group support.
  Arms: Support Group

SUMMARY:
The purpose of this study is to determine whether telephone-adapted Mindfulness Based Stress Reduction (tMBSR) - a program of mindfulness meditation and gentle Hatha yoga delivered mostly by phone, is an effective program to reduce symptoms (anxiety, depression, sleep) and improve quality of life for people waiting for a kidney transplant. Participants will be randomly assigned to tMBSR or to a support group emphasizing communication skills and selecting resources. Both 8-week programs include an initial in-person meeting, 6 weekly teleconference calls, and conclude with an in-person meeting. Participants will complete questionnaires at 3 timepoints over 6 months, and if they receive a transplant, will complete additional questionnaires. Participants will complete sleep diaries and wear Actiwatches (similar to a wristwatch) for one week before programs start, and when programs end, to measure sleep. Participants will provide saliva samples, over 3 days before programs start, and again when programs end, to measure salivary cortisol, an indicator of stress. tMBSR participants will record daily home meditation practice.

DETAILED DESCRIPTION:
Primary Aims

1. Test the efficacy of a telephone-adapted Mindfulness-Based Stress Reduction (tMBSR) program to reduce symptoms and improve the quality of life of kidney transplant candidates by 8-weeks and by 6-month follow-up.
2. Evaluate the impact of tMBSR on sleep measured by actigraphy, and on physiologic stress, as indicated by alteration in the slope of diurnal salivary cortisols, measured before and at the end of the 8-week active intervention period.

Secondary Aims

1. Evaluate the impact of tMBSR on perceptions of transplant surgery (treatment satisfaction, pain) and of Health Related Quality of Life (HRQL) at 2-, 6- and 12-mos post-transplant surgery.
2. Design a full-scale randomized controlled trial (RCT) of the effectiveness and cost-effectiveness of tMBSR.

Hypotheses

* Primary: The tMBSR group will report better outcomes than an attention control support group (SG) on standardized scales for anxiety, depression, and sleep quality and health-related quality of life at 8 weeks and 6 month follow-up.
* Secondary: The tMBSR group will report better outcomes than the SG group on actigraphy-derived sleep parameters and diurnal salivary cortisol patterns.
* Tertiary: Candidates who attended mindfulness training will report greater treatment satisfaction, less distress from pain with transplant surgery and better HRQL 2 months, 6 months and 1 year after kidney transplantation.

Rationale for study : For patients with living with kidney failure, the wait for new kidney is a stressful time. Pharmacologic therapies for managing symptoms of stress increase risks for side effects and non-adherence. Mindfulness-based stress reduction (MBSR), a non-pharmacologic program of training in mindfulness meditation, could help these patients reduce their symptom distress without increasing these other risks.

Long-range Goal: To develop evidence-based recommendations for non-pharmacologic strategies that provide symptom relief to transplant patients, and are safe, practical and cost-effective.

Interventions: The tMBSR program includes the curricular content of the standard 8-week MBSR program (2002 Instructor's Manual). A trained teacher provides instruction in meditation techniques including the body-scan, standing, sitting and walking meditations, and gentle Hatha yoga. Whereas the standard MBSR is conducted as 8 weekly 2.5 hour classes with a one day retreat between weeks 6 and 7, the telephone-adapted MBSR program begins with 5 hour-day workshop to introduce the techniques, followed by 6 weekly 1 ½ hour group teleconferences with the teacher to discuss the class's experiences with meditation practice, and ends with a 5 hour retreat in week 8. Home practice expectations are 25 minutes per day, 6 days a week for tMBSR.

The attention control consists of two 90 minute in-person workshops and 6 1-hour teleconference calls. An experienced facilitator emphasizes communication skills and group support.

Recruiting Methods:

1. Direct mail to candidates being followed by the Transplant Information Services Office with follow-up calls; invitation letters and brochures sent from the P01 Clinical Core.
2. Posters and flyers in medical clinics.
3. Referral by health providers - in- service presentations to the pre-transplant coordinators who manage the kidney candidates;
4. Additional invitations letters mailed by the coordinator who maintains the waitlist for the United Network for Organ Sharing (UNOS); study brochure or invitation letters mailed with waitlist acceptance letters.

Potential Measures of intervention 'dose' or enactment:

1. Mindfulness scale: Mindful Awareness Attention Scale (MAAS);
2. Meditation practice time.

Exploratory Outcomes: Post-transplant impact on Quality of Life (QOL) by Short-Form-36 item(SF-36), pain and satisfaction with transplant hospitalization.

Evaluation Methods:

1. Self-report, mailed questionnaires completed at study weeks 0, 8, 26 (primary outcomes and QOL measures),
2. Actigraphy recording for 1 week prior to the intervention and during the last week of the intervention; cortisol collection for 3 days during same time periods.
3. Post transplant evaluations - 2 and 6 mos; 1 year coordinated with Transplant Database

Duration of Treatment: 8 weeks

Study Duration: Participants are followed up to one year post-kidney transplant.

Statistical Considerations: This study is powered to compare MBSR and SG, on the primary endpoint, on the State Trait Anxiety Inventory (STAI), at 8 weeks. Randomization may be stratified by dialysis (yes/no) and history of diabetes (yes/no).

ELIGIBILITY:
Inclusion Criteria:

* Candidate on the United Network for Organ Sharing (UNOS) wait list for a kidney or kidney-pancreas or evaluated as eligible for candidacy at the UMN
* Aged 18 or older
* English-speaking
* Literate
* Mentally intact
* Able to use the telephone to participate in 6 weekly teleconferences
* Able to attend 2 in-person classes in a Minnesota Metro area
* Able to comply with study monitoring requirements
* Receiving standard medical follow-up care
* Willing to complete the informed consent process

Exclusion Criteria:

* Prior transplant
* Medically unstable (a hospital admission for non-elective purposes in the last 3 months or major non-transplant surgery planned in the next 3 months)
* Serious preexisting mental health issues: suicidality or thought disorder/psychosis; or delirium or substance abuse
* Not expected to be on the waiting list > 3 months (e.g., acceptable living donor has been identified and scheduled)
* Prior MBSR class or regularly practicing mindfulness meditation (twice a week or more)
* Not receiving standard medical care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-02; Primary Completion 2014-06 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia R Gross, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gross CR, Kreitzer MJ, Reilly-Spong M, Winbush NY, Schomaker EK, Thomas W. Mindfulness meditation training to reduce symptom distress in transplant patients: rationale, design, and experience with a recycled waitlist. Clin Trials. 2009 Feb;6(1):76-89. doi: 10.1177/1740774508100982. PMID 19254938
- [Background] Gross CR, Kreitzer MJ, Russas V, Treesak C, Frazier PA, Hertz MI. Mindfulness meditation to reduce symptoms after organ transplant: a pilot study. Altern Ther Health Med. 2004 May-Jun;10(3):58-66. PMID 15154154
- [Background] Kreitzer MJ, Gross CR, Ye X, Russas V, Treesak C. Longitudinal impact of mindfulness meditation on illness burden in solid-organ transplant recipients. Prog Transplant. 2005 Jun;15(2):166-72. doi: 10.1177/152692480501500210. PMID 16013466
- [Background] Kreitzer MJ, Gross CR, Waleekhachonloet OA, Reilly-Spong M, Byrd M. The brief serenity scale: a psychometric analysis of a measure of spirituality and well-being. J Holist Nurs. 2009 Mar;27(1):7-16. doi: 10.1177/0898010108327212. Epub 2009 Jan 28. PMID 19176898
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553
- [Derived] Gross CR, Reilly-Spong M, Park T, Zhao R, Gurvich OV, Ibrahim HN. Telephone-adapted Mindfulness-based Stress Reduction (tMBSR) for patients awaiting kidney transplantation. Contemp Clin Trials. 2017 Jun;57:37-43. doi: 10.1016/j.cct.2017.03.014. Epub 2017 Mar 22. PMID 28342990
- [Derived] Reilly-Spong M, Reibel D, Pearson T, Koppa P, Gross CR. Telephone-adapted mindfulness-based stress reduction (tMBSR) for patients awaiting kidney transplantation: Trial design, rationale and feasibility. Contemp Clin Trials. 2015 May;42:169-84. doi: 10.1016/j.cct.2015.03.013. Epub 2015 Apr 3. PMID 25847578

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 66 people were screened, 3 were ineligible, and of the 63 who consented only 55 actually participated in the trial.
Period: Overall Study
Arm/Group | tMBSR | Support Group
Started | 27 | 28
Completed | 24 | 27
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | tMBSR | Support Group | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 4 | 5 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 31
  Male | 8 | 16 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 2 | 8
  White | 19 | 23 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: State-Trait Anxiety Inventory
Description: The STAI is a 20 item scale that measures current anxiety symptoms with scores that range from 20 to 80, with higher scores indicating greater levels of anxiety. The norm for working adults is a score of 34.
Time Frame: Baseline, 8 weeks, 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tMBSR | Support Group
Number analyzed (Participants) | 24 | 27
units on a scale
  Baseline | 42.1 (12.7) | 37.8 (12.7)
  8 weeks | 40.6 (15.0) | 34.8 (10.0)
  26 weeks | 41.2 (15.3) | 38.1 (11.6)

2. Secondary Outcome: Short Form -12 MCS
Description: Mental component summary score (MCS) of the SF-12 is a self-reported measure of mental health-related quality of life. Scores are reported as standardized T-scores, where an average (mean) score in the general population is 50 with a standard deviation of 10. Scores of 40 or less indicate impaired mental health quality or function.
Time Frame: baseline, 8 and 26 weeks
Measure: Mean (Standard Deviation); unit: T-Scores
Arm/Group | tMBSR | Support Group
Number analyzed (Participants) | 24 | 27
T-Scores
  baseline | 48.9 (8.6) | 49.6 (7.7)
  8 week | 48.3 (8.4) | 51.1 (7.2)
  26 week | 49.7 (9.9) | 46.7 (9.8)

3. Secondary Outcome: SF-12 PCS
Description: Physical component summary score (PCS) of the SF-12 is a self-reported measure of physical health-related quality of life.Scores are reported as standardized T-scores, where an average (mean) score in the general population is 50 with a standard deviation of 10. Scores of 40 or less indicate impaired physical health quality or function.
Time Frame: baseline, 8 weeks, 26 weeks
Measure: Mean (Standard Deviation); unit: T scores
Arm/Group | tMBSR | Support Group
Number analyzed (Participants) | 24 | 27
T scores
  baseline | 34.5 (11.0) | 38.1 (11.0)
  8 week | 38.1 (10.5) | 38.3 (11.3)
  26 week | 33.2 (9.8) | 38.5 (10.4)

4. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI is a 19-item self-reported sleep quality measure with scores that range from 0 to 21, where higher scores indicate worse sleep quality. Scores greater than 5 indicate poor sleep.
Time Frame: baseline, 8 weeks, 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tMBSR | Support Group
Number analyzed (Participants) | 24 | 27
units on a scale
  baseline | 7.4 (3.6) | 6.3 (3.7)
  8 week | 7.3 (4.7) | 6.1 (3.4)
  26 week | 8.5 (5.4) | 7.1 (4.1)

5. Secondary Outcome: Center for Epidemiologic Studies Depression Scale (CESD)
Description: The CES-D is a 20-item self-report scale to measure symptoms of depression in the past week with scores having a range of 0 to 60 and a score of 16 or higher indicating clinically relevant symptoms.
Time Frame: baseline, 8 weeks, 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tMBSR | Support Group
Number analyzed (Participants) | 24 | 27
units on a scale
  baseline | 15.4 (9.9) | 11.1 (7.5)
  8 week | 14.7 (9.4) | 9.1 (5.8)
  26 week | 16.9 (11.6) | 11.1 (8.6)

ADVERSE EVENTS:
Arm/Group | tMBSR | Support Group
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 0/27 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No